CLINICAL TRIAL: NCT02590731
Title: The Influence of Cognitive Status on Walking Abilities After Hemiarthroplasty for Femoral Neck Fracture: a Prospective Cohort Study
Brief Title: The Influence of Cognitive Status on Walking Abilities After Femoral Neck Fracture
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SM_III
Record Dates: First submitted 2015-10-13; First posted 2015-10-29 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Hip Fracture; Femoral Neck Fracture
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Pfeiffer test 6 or above. No or mild cognitive impairment
- Cognitivt impaired: Pfeiffer test less than 6. Moderate to severe cognitive impairment.

SUMMARY:
Introduction: Femoral neck fracture is a devastating injury with serious medical and social consequences. One third of these patients have some degree of impaired cognitive status. Despite of this, a high proportion of hip fracture trials exclude patients with cognitive impairment. The investigators aimed to evaluate whether moderate to severe cognitive impairment could predict walking ability, quality of life, functional outcome, reoperations and mortality in elderly patients treated with hemiarthroplasty.

Methods: This cohort study included a consecutive series of 188 patients treated with hemiarthroplasty for an displaced femoral neck fracture. Patient were assessed for estimated preoperative and 1 year postoperatively with regard to walking abilities, cognitive status, quality of life with EQ-5D and hip function with Harris hip score.

ELIGIBILITY:
Inclusion Criteria:

* 65 year or above
* Displaced femoral neck fracture
* Treated with a hemiarthroplasty

Exclusion Criteria:

* Pathological fractures
* Bilateral femoral neck fractures
* Bed-ridden patients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient with displaced femoral neck fractures.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Walking abilities | 2 years
  At follow-up patients report whether they are walking or not by questionnaire

SECONDARY OUTCOMES:
Harris hip score | 2 years
EQ-5D | 2 years
Reoperation | 2 years
Mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mukka, M.D, PhD, Principal Investigator — Umeå University

REFERENCES:
- [Background] Hedbeck CJ, Inngul C, Blomfeldt R, Ponzer S, Tornkvist H, Enocson A. Internal fixation versus cemented hemiarthroplasty for displaced femoral neck fractures in patients with severe cognitive dysfunction: a randomized controlled trial. J Orthop Trauma. 2013 Dec;27(12):690-5. doi: 10.1097/BOT.0b013e318291f544. PMID 23515127